CLINICAL TRIAL: NCT04710732
Title: Individual Dose Adjustment of Low-molecular-weight-heparin by Thromodynamics Test in Patients At Extremely High Risk of Postoperative Venous Thromboembolism.
Brief Title: Individual Dose Adjustment of Low-molecular-weight-heparin by Thromodynamics Test.
Acronym: IDAHeT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of the eligible patients
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Kirill Lobastov, Associate Professor, Pirogov Russian National Research Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IDAHeT
Record Dates: First submitted 2021-01-09; First posted 2021-01-15 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Venous Thromboembolism
Keywords: deep vein thrombosis; pulmonary embolism; venous thromboembolism; caprini score; prophylaxis; low molecular weight heparin
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): Peri-operative VTE prophylaxis with a standard once-daily dose of enoxaparin 40 mg and anti-embolic stockings
  Interventions: Drug: Standard Enoxaparin 40 mg once-daily before randomization; Drug: Standard Enoxaparin 40 mg once-daily after randomization; Device: Anti-embolic elastic compression stockings; Diagnostic Test: Thrombodynamic test (TD)
- Experimental (Experimental): Peri-operative VTE prophylaxis with an escalated twice-daily dose of enoxaparin 30 mg and anti-embolic stockings
  Interventions: Drug: Standard Enoxaparin 40 mg once-daily before randomization; Drug: Escalated Enoxaparin 30 mg twice-daily after randomization; Device: Anti-embolic elastic compression stockings; Diagnostic Test: Thrombodynamic test (TD)

INTERVENTIONS:
Drug: Standard Enoxaparin 40 mg once-daily before randomization — Once-daily subcutaneous injection of a standard prophylactic dose of Enoxaparin 40 mg according to the set schedule:
  * 12 hours before the surgery (if applicable) on a postoperative day -1 (POD -1)
  * 6-12 hours after the surgery (key injection 1) on the surgery day (POD 0)
  * 12 hours after the previous key injection 1 (key injection 2) on the POD 1
  * 24 hours after the previous key injection 2 on the POD 2
Drug: Standard Enoxaparin 40 mg once-daily after randomization — Once-daily subcutaneous injection (every 24 hours) of a standard prophylactic dose of Enoxaparin 40 mg since POD 3 and until discharge
  Arms: Control
Drug: Escalated Enoxaparin 30 mg twice-daily after randomization — Twice-daily subcutaneous injection (every 12 hours) of an escalated prophylactic dose of Enoxaparin 30 mg since POD 3 and until discharge
  Arms: Experimental
Device: Anti-embolic elastic compression stockings — Applied before or just after the surgery and used around the clock until discharge
Diagnostic Test: Thrombodynamic test (TD) — Blood sampling for TD:
  * 12 hours after key injection 1 (TD-12) on the POD 1
  * 24 hours after key injection 2 (TD-24) on the POD 2
  * 24 hours after each daily injection on the POD 4 (TD-4) and POD 5 (TD-5)

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of individual dose adjustment of low molecular weight heparin (LMWH) based on the results of the thrombodynamics test (TD) in patients at extremely high risk of postoperative venous thromboembolism (VTE).

This is a single-center, open-label, randomized clinical study with a blinded assessor for primary efficacy outcome.

Patients after elective or emergent major surgery having 10 or more Caprini scores at the baseline, who already received two subcutaneous injections of enoxaparin: 40 mg at 6-12 hours after the surgery ("key injection 1") and 40 mg at 12 hours after the previous injection ("key injection 2"), who had no VTE at the baseline, and who signed informed consent, are subjected to laboratory examination by the TD.

Blood samples are taken 12 hours after the "key injection 1" and 24 hours after the "key injection 2". If one of the relevant parameters of the TD (initial velocity of clot growth rate and clot size) exceeds the set threshold, the Caprini scores are recalculated adding 3 points for "other thrombophilic state" confirmed by the thrombodynamics. The patient may be included in the study if the new sum exceeds 13 points (initial 10 scores + additional 3 scores). Within 60 hours from the surgery, the included patients are randomly allocated to one of two groups: Experimental or Control. Patients in the Control group continue to receive the standard dose of enoxaparin 40 mg every 24 hours (once daily). In the Experimental group, the dose of enoxaparin is increased to 30 mg every 12 hours (twice daily).

Blood samples for TD are taken during the next two days at 24 hours after the administration of each daily dose of enoxaparin.

A whole leg duplex ultrasound scan (DUS) is performed in all patients during the screening period and at 7-10 days after the surgery or in case of any suspicion for deep vein thrombosis (DVT) or superficial vein thrombosis (SVT). Computed tomography pulmonary angiography (CTPA) is carried out in any clinical suspicion for pulmonary embolism (PE). An autopsy is performed in all dead patients.

The total follow-up period is 30 days. After discharge, patients are invited to the hospital for clinical examination with DUS or interviewed by phone to identify symptomatic VTE.

ELIGIBILITY:
Inclusion Criteria:

* performed major surgery;
* performed the key injection 1 and the key injection 2 of enoxaparin 40 mg;
* performed thrombodynamics test at 12 hours after the key injection 1 and at 24 hours after the key injection 2;
* at least one of the relevant TD parameters exceeds the set threshold: initial velocity of clot growth >62.5 μm / min at 12 hours after the key injection 1, or initial velocity of clot growth >64.5 μm / min at 24 hours after the key injection 2, or clot size >1333.5 μm at 12 hours after the key injection 1, or clot size >1351.5 μm at 24 hours after the key injection 2;
* Caprini score of 13 and higher after recalculation with the results of the TD test;
* infirmed consent is given.

Exclusion Criteria:

* 60 or more hours passed since the end of surgery;
* venous thrombosis at the baseline;
* performed partial occlusion of the inferior vena cava (plication, filter);
* indications for the use of anticoagulants in different regimen;
* high risk of bleeding;
* contraindication to anticoagulation;
* contraindication to elastic compression;
* inability for blood sampling from a peripheral vein;
* anticipated death within 5 days or less.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Symptomatic and asymptomatic venous thrombosis by postoperative day 10 | day 10 after surgery
  The number of patients with a combination of asymptomatic DVT or SVT revealed by routine DUS performed by blinded assessor between 7 and 10 postoperative day and symptomatic DVT or SVT confirmed by unscheduled DUS.

SECONDARY OUTCOMES:
The number of patients with the reduction of any relevant parameter of the TD test by postoperative day 5 | day 5 after surgery
  The number of patients in whom any relevant parameter of the TD test does not exceed the set threshold at control blood test on POD-5 (TD-5):
  -initial velocity of clot growth (Vin) <62.5 μm / min at 12 hours after enoxaparin 30 mg injection (experimental group) or <64.5 μm / min at 24 hours after enoxaparin 40 mg injection (control group)
  or
  -clot size (CS): <1333.5 μm at 12 hours after enoxaparin 30 mg injection (experimental group) or <1351.5 μm / min at 24 hours after enoxaparin 40 mg injection (control group)
The number of patients with the reduction of all relevant parameters of the TD test by postoperative day 5 | day 5 after surgery
  The number of patients in whom all relevant parameters of the TD test do not exceed the set threshold at control blood test on POD-5 (TD-5):
  -initial velocity of clot growth (Vin) <62.5 μm / min at 12 hours after enoxaparin 30 mg injection (experimental group) and <64.5 μm / min at 24 hours after enoxaparin 40 mg injection (control group)
  and
  -clot size (CS): <1333.5 μm at 12 hours after enoxaparin 30 mg injection (experimental group) and <1351.5 μm / min at 24 hours after enoxaparin 40 mg injection (control group)
The number of patients with the normalization of every parameter of the TD test by postoperative day 5 | day 5 after surgery
  The number of patients in whom every parameter of the TD test does not exceed the upper limit of normal at control blood test on POD-5 (TD-5):
  * initial velocity of clot growth (Vin) <56 μm / min, and
  * clot size (CS): <1200 μm, and
  * lag-time: >0.6 sec, and
  * stationary velocity of clot growth: <29 μm / min, and
  * clot density: <32000 c.u., and
  * spontaneous clots: negative.
Symptomatic and asymptomatic venous thromboembolism by postoperative day 10 | day 10 after surgery
  The number of patients with a combination of asymptomatic DVT or SVT revealed by routine DUS performed by blinded assessor between 7 and 10 postoperative day and symptomatic DVT, SVT, or PE confirmed by unscheduled DUS, CTPA, or autopsy.
Symptomatic pulmonary embolism by postoperative day 10 | day 10 after surgery
  The number of patients with symptomatic pulmonary embolism confirmed by CTPA or autopsy
Fatal pulmonary embolism by postoperative day 10 | day 10 after surgery
  The number of patients with fatal pulmonary embolism confirmed by autopsy
Death by postoperative day 10 | day 10 after surgery
  The number of patients who died for any reason within 10 days after surgery
Symptomatic and asymptomatic venous thromboembolism by postoperative day 30 | day 30 after surgery
  The number of patients with a combination of asymptomatic DVT or SVT revealed by routine DUS performed by blinded assessor between 7 and 10 postoperative day and symptomatic DVT, SVT, or PE confirmed by appropriate medical image or autopsy within 30 days after surgery as revealed by clinical examination, the examination of medical records or telephone interview.
Death by postoperative day 30 | day 30 after surgery
  The number of patients who died for any reason within 30 days after surgery as revealed by the telephone interview and/or examination of medical records.
Major bleeding by postoperative day 30 | day 30 after surgery
  The number of patients with major bleeding as defined by the International Society of Thrombosis and Hemostasis occurred within 30 days after surgery as assessed by the Data Monitoring Committee.
Clinically relevant non-major bleeding by postoperative day 30 | day 30 after surgery
  The number of patients with clinically relevant non-major bleeding as defined by the International Society of Thrombosis and Hemostasis occurred within 30 days after surgery as assessed by the Data Monitoring Committee.
Minor bleeding by postoperative day 30 | day 30 after surgery
  The number of patients with any other bleeding not fulfilling the criteria of major nor clinically relevant non-major bleeding that occurred within 30 days after surgery as assessed by the Data Monitoring Committee.

CONTACTS AND LOCATIONS:
Overall Officials: Kirill Lobastov, PhD, Principal Investigator — Pirogov RNRMU
Locations (1):
- Moscow Clinical Hospital no.24, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided